CLINICAL TRIAL: NCT02059343
Title: Pharmacokinetics of Dexmedetomidine in Children During Cardiopulmonary Bypass (CPB)
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00049942; K24HD05873505 (Other Grant/Funding Number: NICHD)
Record Dates: First submitted 2014-02-05; First posted 2014-02-11 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-10

CONDITIONS: Pharmacokinetics; Cardiopulmonary Bypass; Children
Keywords: pharmacokinetics; pharmacodynamics; safety; dexmedetomidine; cardiopulmonary bypass; children

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood will be collected for plasma pharmacokinetic analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- age less than or equal to 2 years

SUMMARY:
Dexmedetomidine is increasingly used for sedation in children placed on cardiopulmonary bypass for heart surgery. It is also often used after surgery and may be particularly helpful for children with heart disease. In order for this medication to be helpful and to minimize risks associated with taking the medication, it is important to provide correct dosing for this medication. Based on evidence from studies of other medications used during heart surgery, it is likely that dosing of dexmedetomidine while on cardiopulmonary bypass is different from dosing in other settings. The purpose of this study is to evaluate how the heart-lung bypass machine affects dexmedetomidine levels in the body.

ELIGIBILITY:
Inclusion Criteria:

* < 2 years of age
* Sufficient venous access to permit administration of study medication.
* Supported with cardiopulmonary bypass (CPB)
* Receiving dexmedetomidine per standard of care.
* Availability and willingness of the parent/legal guardian to provide written informed consent.

Exclusion Criteria:

* <38 weeks post menstrual age
* Any concomitant condition, which in the opinion of the investigator would preclude a subject's participation in the study.
* Previous participation in this study
* CPB circuit primed with clear fluid

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will include children less than or equal to 2 years of age who undergo cardiopulmonary bypass and receive dexmedetomidine per standard of care during the bypass session.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2014-03; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetics (clearance, volume of distribution, area under the curve, oxygenator extraction efficiency) of dexmedetomidine in children supported with cardiopulmonary bypass | Data will be collected at the following approximate time points: 0h, 0.5h, 0.75h, and 2h after infusion initiation; 0.25h, 0.75h, and 2h after bypass initiation; 0.5h prior to bypass termination, 0.25h, 1h, 3h, 7h, and 10h after bypass termination
  The plasma pharmacokinetics of dexmedetomidine will include
  * Clearance (CL)
  * Volume of distribution (V)
  * Area under the curve (AUC)
  * Oxygenator extraction efficiency

SECONDARY OUTCOMES:
COMFORT behavioral score as a measure of dexmedetomidine pharmacodynamics | assessed at time 0, upon presentation to the intensive care unit after surgery, and 12-24 hours from study drug initiation.
Accessory sedative and analgesic use as a measure of dexmedetomidine pharmacodynamics | up to 48 hours after study drug initiation
  We will monitor sedatives and analgesics used in addition to dexmedetomidine. Quantification of use of other drugs will allow an indication of the sedative effects of dexmedetomidine.

OTHER OUTCOMES:
Vital sign variation as a measure of safety | up to 48 hours after study drug initiation
  Adverse events of special interest will be evaluated. These will include the presence of bradycardia, hypertension, and hypotension that occur after administration of dexmedetomidine

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Watt, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States